CLINICAL TRIAL: NCT07251764
Title: Study of the Blood-Interstitial Glucose Gap and Its Prediction of Metabolism and Prognosis in Critically Ill Patients
Brief Title: The Blood-Interstitial Glucose Gap
Status: Completed | Type: Observational
Sponsor: Chinese Medical Association (Network)
Responsible Party: Sponsor
Other Study IDs: Zhibo Zhang
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Critical Illness; Metabolism Disorders
Keywords: Glucose Gap; Metabolic Monitoring; Prognosis; Insulin Resistance
MeSH Terms: conditions — Critical Illness; Metabolic Diseases; Insulin Resistance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Metabolic monitoring is fundamental to guiding nutritional therapy in critically ill patients. Although indirect calorimetry is the established gold standard for measuring resting energy expenditure, its routine clinical use is constrained by practical challenges, including procedural complexity, time-intensive nature, significant cost, and limited feasibility in patients on advanced life support, such as extracorporeal membrane oxygenation (ECMO). Dysregulation of glucose metabolism is common in this population, characterized not only by absolute dysglycemia but also-and perhaps more critically-by impairments in the efficiency of glucose transport and utilization across the microcirculatory continuum (from arterial blood, through the interstitial space, to venous return). This study seeks to examine the relationship between novel dynamic metrics-such as the arterio-interstitial glucose gradient-and key clinical parameters, including energy expenditure, organ function, and patient outcomes. Our objective is to assess the utility of these measures as minimally invasive, real-time biomarkers of metabolic state in critical illness.

DETAILED DESCRIPTION:
This prospective observational study aims to investigate the association between blood-interstitial fluid glucose concentration differences and resting energy expenditure, organ function, and clinical outcomes in critically ill patients, while also exploring potential factors influencing these glucose concentration differences.

ELIGIBILITY:
Inclusion Criteria:

* Age≥ 18 years and < 80 years
* ICU stay ≤48 hours
* Expected ICU stay > 24 hours
* APACHE II score≥ 8

Exclusion Criteria:

* local infection within the sensor placement area
* Laparotomy within lower abdomen
* Participated in this study before
* In other clinical trails

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: critically ill patient
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2023-07-13 (Actual); Primary Completion 2024-03-13 (Actual); Study Completion 2025-10-01 (Actual)

PRIMARY OUTCOMES:
ICU Mortality | From date of study enrollment until the date of ICU discharge or date of death from any cause, whichever came first, assessed up to 60 days
  The incidence of all-cause death during the patient's stay in the Intensive Care Unit

SECONDARY OUTCOMES:
Duration of Vasopressor Dependency | From date of study enrollment until the date of vasopressor cessation for at least 24 hours, assessed up to 30 days
  The total length of time a patient requires continuous intravenous vasoactive drugs to maintain adequate blood pressure.
Duration of Invasive Mechanical Ventilation | From date of study enrollment until the date of successful extubation, tracheostomy, or death from any cause, whichever came first, assessed up to 30 days
  The total length of time a patient requires endotracheal intubation and support from a mechanical ventilator.
Duration of Continuous Renal Replacement Therapy (CRRT) | From date of study enrollment until the date of CRRT discontinuation for at least 24 hours or death from any cause, whichever came first, assessed up to 30 days
  The total length of time a patient requires continuous renal replacement therapy for acute kidney injury.

CONTACTS AND LOCATIONS:
Overall Officials: Wenkui Yu, Professor, Principal Investigator — The Affiliated Nanjing Drum Tower Hospital of Nanjing University Medical School
Locations (1):
- Nanjing Drum Tower Hospital, Nanjing, Jiangsu, China